CLINICAL TRIAL: NCT03069950
Title: A Randomized, Multicenter Phase II Study of Panitumumab Plus FOLFIRI With or Without Hepatic Arterial Infusion as Second-Line Treatment in Patients With Wild Type RAS Who Have Unresectable Hepatic Metastases From Colorectal Cancer
Brief Title: Study of Chemotherapy With or Without Hepatic Arterial Infusion for Patients With Unresectable Metastatic Colorectal Cancer to the Liver
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The Cleveland Clinic (Other); Oregon Health and Science University (Other); Queens Cancer Center of Queens Hospital (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1341
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Adenocarcinoma Metastatic to the Liver
Keywords: Hepatic Arterial Infusion; Floxuridine (FUDR); Irinotecan (CPT-11); FLUOROURACIL; PANITUMUMAB; 16-1341
MeSH Terms: interventions — Floxuridine; Irinotecan; Fluorouracil; Panitumumab; Dexamethasone; Leucovorin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HAI FUDR/Dex in addition to Pmab plus FOLFIRI (Experimental): Panitumumab plus FOLFIRI on Day 1 and Day 15 of each cycle. HAI pump therapy with FUDR and Dex on Day 1 of each cycle. Patients will start protocol therapy approximately 2 weeks after surgery. All patients will receive Panitumumab (6 mg/kg IV over 60 min). The HAI FUDR group will receive FOLFIRI in the following dosing; 5-Fluouracil (5FU) (1000 mg/m2/day continuous infusion over two days), Leucovorin (LV) (400 mg/m2 IV over 30 min to an hour), and Irinotecan (CPT) (150 mg/m2 IV over 30 min to an hour) on Day 1 and Day 15.
  Interventions: Drug: Floxuridine (FUDR); Drug: Irinotecan (CPT-11); Drug: FLUOROURACIL; Drug: PANITUMUMAB; Drug: DEXAMETHASONE; Drug: Leucovorin
- Pmab plus FOLFIRI alone (Experimental): The dosing of FOLFIRI in the systemic arm will be 5-Fluouracil (5FU) (1200 mg/m2/day continuous infusion over two days), Leucovorin (LV) (400 mg/m2 IV over 30 min to an hour), bolus 5FU 400mg/ m2 and Irinotecan (CPT) (150 mg/m2 IV over 30 min to an hour) on Day 1 and 15.
  Interventions: Drug: Floxuridine (FUDR); Drug: Irinotecan (CPT-11); Drug: FLUOROURACIL; Drug: PANITUMUMAB; Drug: Leucovorin

INTERVENTIONS:
Drug: Floxuridine (FUDR) — 5-Fluouracil (5FU) (1000 mg/m2/day continuous infusion over two days)
Drug: Irinotecan (CPT-11) — Irinotecan (CPT) (150 mg/m2 IV over 30 min to an hour) on Day 1 and Day 15.
Drug: FLUOROURACIL — 5-Fluouracil (5FU) (1200 mg/m2/day continuous infusion over two days)
Drug: PANITUMUMAB — Panitumumab (6 mg/kg IV over 60 min)
Drug: DEXAMETHASONE — flat dose of 25 mg on Day 1
  Arms: HAI FUDR/Dex in addition to Pmab plus FOLFIRI
Drug: Leucovorin — Leucovorin (LV) (400 mg/m2 IV over 30 min to an hour)

SUMMARY:
The purpose of this study is to see if patients treated with both regional chemotherapy using the HAI pump and intravenous chemotherapy are able to have their liver tumors removed surgically (resected), versus treatment with only intravenous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed colorectal adenocarcinoma metastatic to the liver with no clinical or radiographic evidence of extrahepatic disease. Confirmation of diagnosis must be performed by the enrolling institution.
* Patients must have a primary L sided colorectal cancer, (at or distal to the splenic flexure)
* Confirmed RAS/RAF wild type tumor. Paraffin-embedded tumor tissue obtained from the primary tumor or metastasis
* Have received prior treatment for metastatic disease with oxaliplatin-based regimen and either

  * Had disease progression OR
  * Had stable disease OR
  * Discontinued oxaliplatin due to neuropathy
* Patients must meet the following criteria for unresectability as determined by two hepatobiliary surgeons and one radiologist:

  * When a margin negative resection would require resection of all three hepatic veins, both portal veins, or the retrohepatic vena cava.
  * Requiring a resection that leaves less than 2 hepatic segments (not including the caudate lobe) behind with adequate arterial/portal inflow, venous outflow and biliary drainage. **

    **A patient is considered resectable if the procedure includes a minor wedge or thermo-ablation encompassing 10% or less of the volume of the remaining 2 segments.
  * Patient"s liver metastases must comprise <70% of the liver parenchyma. All patients must be clinically fit to undergo surgery as determined by the pre-operative evaluation
* Lab values within 14 days prior to enrollment/randomization:

  * WBC ≥ 3.0 K/uL
  * ANC > 1.5 K/uL
  * Platelets ≥ 100,000/uL
* Renal function (≤ 10 days prior to enrollment/randomization) °Creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min calculated by the Cockcroft-Gault method as follows:

Cockcroft-Gault method as follows:

* Male creatinine clearance = (140 -age in years) x (weight in Kg) / (serum Cr in mg/dl x 72)
* Female creatinine clearance = (140 - age in years) x (weight in Kg) x 0.85 / (serum Cr in mg/dl x 72) (use of creatinine clearance per protocol based on chemotherapy regimen)

  * Hepatic function, as follows: (≤ 10 days prior to enrollment/randomization)
* Total Bilirubin ≤ 1.5 mg/dl

  * Calcium ≥ lower limit of normal (≤ 48 hours prior to enrollment/randomization)
  * KPS ≥ 60% (ECOG (or Karnofsky) performance status (preferably 0 or 1/≥ 60% for Karnofsky))

Exclusion Criteria:

* Patients < 18 years of age
* Patients who have received more than one chemotherapy regimen for metastatic disease
* Patients who are chemotherapy naïve
* Prior radiation to the liver (Prior radiation therapy to the pelvis is acceptable if completed at least 4 weeks prior to registration)
* Active infection

  °Active infection includes patients with positive blood cultures
* Prior treatment with HAI FUDR
* Prior TACE
* Female patients who are pregnant or lactating - or planning to become pregnant within 6 months after the end of the treatment (female patients of child-bearing potential must have negative pregnancy test ≤ 72 hours before enrollment and randomization, and must have a negative pregnancy test ≤ 72 hours prior to treatment start)
* If a patient has any serious medical problems which may preclude receiving this type of treatment
* Patients with history or known presence of primary CNS tumors, seizures not well-controlled with standard medical therapy, or history of stroke will also be excluded.
* Serious or non-healing active wound, ulcer, or bone fracture
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Patients who have a diagnosis of Gilbert"s disease
* History of other malignancy, except:

  1. Malignancy treated with curative intent and with no known active disease present for ≥ 3 years prior to randomization and felt to be at low risk for recurrence by the treating physician
  2. Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated cervical carcinoma in situ without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Resection rate assessed using RECIST (version 1.1) | 3 months
  Treatment evaluation will be done using RECIST (version 1.1) The patient will be assessed with repeat CT scans as specified. If at any time after 3 cycles (or 3 months) the patient is able to undergo a complete resection of all hepatic metastases they will proceed to operative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memoral Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm